CLINICAL TRIAL: NCT01205516
Title: Methadone in Neuropathic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding agency withdrew funding due to slow recruitment
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Nova Scotia Health Research Foundation (Other Government); Dalhousie University (Other)
Responsible Party: Principal Investigator, Mary Lynch, MD FRCPC, Nova Scotia Health Authority
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDHA-RS/2010-Meth
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2017-07

CONDITIONS: Chronic Neuropathic Pain
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Experimental)
  Interventions: Drug: Methadone
- Controlled Release Morphine (Active Comparator): Controlled release morphine supplied in 10 mg tablets, 1-12 tablets taken twice daily, every 12 hours (range 20-240 mg per 24 hours).
  Interventions: Drug: Controlled Release Morphine

INTERVENTIONS:
Drug: Methadone — Patients in the methadone arm will be supplied with 2.5 mg tablets. The dose will consist of 1-12 tablets taken twice daily, every 12 hours (range 5-60 mg per 24 hours).
  Arms: Methadone
Drug: Controlled Release Morphine — controlled release morphine supplied in 10 mg tablets, 1-12 tablets taken twice daily, every 12 hours (range 20-240 mg per 24 hours).
  Arms: Controlled Release Morphine

SUMMARY:
INTRODUCTION: There is an important need for inexpensive drugs that treat neuropathic pain. Early research suggests that methadone may be a good, inexpensive drug to treat neuropathic pain. Methadone is available in a low cost powder that is easily prepared for different routes of administration. This study will look at the effect and safety of methadone compared to the regular treatment of morphine for the treatment of chronic neuropathic pain.

OBJECTIVES: First the investigators want to determine if methadone is effective and safe for the treatment of neuropathic pain. Since a placebo control group would be unethical, the proposed comparator will consist of the "gold standard" conventional treatment, controlled release morphine. The investigators will compare methadone to controlled-release morphine with regard to how it affects the level of pain and extent of side effects. Next the investigators want to examine safety as well as to determine whether methadone leads to improvements in physical and emotional functioning, and participants' satisfaction with the treatment.

METHODS: A double blind, randomized trial comparing methadone and controlled release morphine is proposed. After 1-week, participants will be randomly assigned to either methadone or controlled release morphine and will gradually build to a dose at which they receive adequate pain relief without unacceptable levels of side effects. This 5-week phase will be followed by a 6-week dose phase and then a 4-week tapering off phase.

Study drug: The study drug is methadone supplied in 2.5 mg tablets. The comparator will consist of controlled release morphine in 10 mg tablets. The dose of each will range from 1-12 tablets taken every 12 hours (dose ranges methadone 5-60 mg/day, controlled release morphine 20-240 mg/day).

Setting: This is a 3-site study involving pain clinics in Halifax, Nova Scotia; London, Ontario; and Calgary, Alberta.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than18 years
* Chronic neuropathic pain of central or peripheral origin for 3 months or longer as determined by the study physician and a score of 4/10 or greater on the DN4
* Moderate to severe pain as defined by average 7-day pain score of greater than 4 on an 11-point numerical rating scale for pain intensity (NRS-PI).
* Physician has identified that an opioid is a valid adjunctive treatment for the chronic neuropathic pain.
* Concomitant non-opioid analgesic medications must have been stable for 14 days.
* Co-interventions such as TENS, acupuncture and massage must have been stable for 14 days prior to the trial
* If taking an opioid, maximum dose of opioid in oral morphine equivalents (OME) is 90 mg/24 hours.
* Ability to follow the protocol with reference to cognitive and situational conditions; e.g., stable housing, able to attend follow-up visits.
* Willing and able to give written informed consent.

Exclusion Criteria:

* Patients on a dose of opioid that exceeds 90 mg/24 hours in OME
* Pregnant or lactating women (women of childbearing potential must have negative pregnancy test)
* History of psychosis
* History of (within the past 2 years) , or current, substance dependency disorder
* Excluded medications are listed in Appendix 1.
* Presence of clinically significant cardiac or pulmonary disorder on physical exam that would compromise participants' safety in the trial as judged by the study physician.
* Presence of significant conduction delay, ischemia or arrhythmia on screening ECG
* Presence of severe pain disorder other than the chronic neuropathic pain under study that would interfere with patient's ability to determine effect of study treatment on the chronic neuropathic pain
* Abnormalities above 1.5 times upper range of normal on screening CBC, blood chemistry including BUN, Cr, LDH, AST, ALT
* Patients with a history of allergy to any opioid.
* Participation in another clinical trial in the 30 days prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
to determine if methadone is an effective opioid for the treatment of chronic neuropathic pain | 16 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - QEII Health Science Centre Pain Management Unit, Halifax, Nova Scotia
  - St. Joseph's Health Care Centre, Neuropathic Pain Clinic, London, Ontario
  - Alan Edwards Pain Management Unit, McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Result] Lynch M, Moulin D, Perez J. Methadone vs. morphine SR for treatment of neuropathic pain: A randomized controlled trial and the challenges in recruitment. Can J Pain. 2019 Oct 22;3(1):180-189. doi: 10.1080/24740527.2019.1660575. eCollection 2019. PMID 35005408